CLINICAL TRIAL: NCT06354556
Title: Effect of Verapamil on the Pharmacokinetic of HRS-1893 Tablets in Healthy Subjects: a Single Center, Open, Single Arm, and Fixed Sequence Study
Brief Title: Effect of Verapamil Tablets on the Pharmacokinetic of HRS-1893 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1893-102
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Verapamil

STUDY DESIGN:
Intervention Model Description: Single center, open, single arm, fixed sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: HRS-1893 tablet; Drug: Verapamil tablet

INTERVENTIONS:
Drug: HRS-1893 tablet — HRS-1893 tablet single dose
Drug: Verapamil tablet — Verapamil tablet 80 mg tid

SUMMARY:
The purpose of this phase Ⅰ study is to evaluate the effect of oral verapamil tablets on the pharmacokinetics of HRS-1893 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in the study, comply with study requirements, and sign the written informed consent form (ICF).
2. Male or female aged 18-55（adult healthy volunteers).
3. Body mass index (BMI) between 19 and 28 kg/m2.
4. Normal Electrocardiogram (ECG).

Exclusion Criteria:

1. History of persistent tachyarrhythmia and syncope.
2. A history of stomach or bowel surgery or excision.
3. Positive results of hepatitis B surface antigen, hepatitis C antibody, syphilis antibody and human immunodeficiency virus antibody.
4. Those who have participated in any clinical trials and have taken study drugs within 3 months before the first administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) for HRS-1893 after Single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Area under the plasma concentration versus time curve from time zero to last measurable timepoint (AUC0-t) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Area under the plasma concentration versus time curve from time zero extrapolated to infinity (AUC0-inf) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (Tmax) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Elimination half-life (T1/2) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Apparent oral clearance (CL/F) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Apparent volume of distribution (Vz/F) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Accumulated amount of excretion (Ae) for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Urinary excretion fraction（fe）for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Renal clearance（CLr）for HRS-1893 after single dose | from Day 1 to Day 8 after the first dose and from Day 12 to Day 19 after the second dose
Number of subjects with adverse events and the severity of adverse events | from Day 1 to Day 24 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided